CLINICAL TRIAL: NCT02566265
Title: Study of High-dose Influenza Vaccine Efficacy by Repeated Dosing IN Gammopathy Patients (SHIVERING 2)
Brief Title: Study of High-dose Influenza Vaccine Efficacy by Repeated Dosing IN Gammopathy Patients
Acronym: SHIVERING 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1507016111
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Influenza; Multiple Myeloma; Waldenstrom's Macroglobulinemia; Plasma Cell Disorders; MGUS
Keywords: influenza; multiple myeloma; Waldenstrom's macroglobulinemia
MeSH Terms: conditions — Influenza, Human; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone High Dose Vaccine then Fluzone High Dose Booster (Experimental): Fluzone High dose vaccine administered at Day 0. Fluzone High dose vaccine administered as a booster after 30 days from the initial vaccine.
  Interventions: Biological: Fluzone High Dose Vaccine
- Standard of Care (Active Comparator): Fluzone High-Dose if age greater than or equal to 65 or Standard dose influenza vaccine if age less than 65 at day 0. Placebo administered 30 days after the initial vaccine.
  Interventions: Biological: Standard of care/Placebo

INTERVENTIONS:
Biological: Fluzone High Dose Vaccine
  Arms: Fluzone High Dose Vaccine then Fluzone High Dose Booster
Biological: Standard of care/Placebo
  Arms: Standard of Care

SUMMARY:
The investigators' hypothesis is that the administration of Fluzone® High-Dose with booster to all patients with monoclonal gammopathies (irrespective of age) will lead to seroconversion rates exceeding 50% and more importantly, will reduce influenza-related morbidity, reduce interruptions in cancer therapy and may reduce disease progression at the end of the flu season

DETAILED DESCRIPTION:
Influenza is a major cause of morbidity in the US. Patients with monoclonal gammopathies are known to have increased risk of developing influenza. Furthermore, several of the medications (such as proteasome inhibitors), commonly used to treat these tumors, are known to further increase the risk of these tumors. Seasonal influenza vaccination has been shown to reduce influenza related morbidity and is approved for routine prophylaxis in US. In 2009, Fluzone® high- dose vaccine was FDA approved in 2009 for adults aged 65 and older based on the data regarding higher rates of seroprotection (defined as hemagglutination antibody inhibition (HAI) titer of 40 or higher).

In this study, the investigators will administer Fluzone® High-Dose vaccine with a planned booster to patients with monoclonal gammopathies irrespective of age versus a standard of care control group. Primary endpoint is composite of documented influenza infection rate and disease progression (as defined by International Myeloma Working Group criteria) at the end of the flu season. Based on the background data, the investigators expect a higher rate of success in the experimental arm. As such, the investigators power for success rates of 90% and 70% in the experimental and control arms, respectively.

The investigators will also analyze several secondary endpoints including rates of influenza related morbidity, the analysis of humoral and cellular immune response to these vaccines and the rate of disease control (defined as lack of disease progression by standard international myeloma working group criteria).

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age ≥18 years at the time of signing the informed consent form.
* Diagnosis of any monoclonal gammopathy: Monoclonal Gammopathy of Undetermined Significance (MGUS), asymptomatic / active multiple myeloma, asymptomatic / active Waldenstrӧm Macroglobulinemia (WM).

Exclusion Criteria:

* Any serious egg allergy or prior serious adverse reaction to an influenza vaccine.
* Use of any other influenza vaccine for the 2015 to 2016 flu season.
* Women who are pregnant or plan to become pregnant in the study period.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-09; Primary Completion 2017-10 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Branagan, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Branagan AR, Duffy E, Gan G, Li F, Foster C, Verma R, Zhang L, Parker TL, Seropian S, Cooper DL, Brandt D, Kortmansky J, Witt D, Ferencz TM, Dhodapkar KM, Dhodapkar MV. Tandem high-dose influenza vaccination is associated with more durable serologic immunity in patients with plasma cell dyscrasias. Blood Adv. 2021 Mar 9;5(5):1535-1539. doi: 10.1182/bloodadvances.2020003880. PMID 33683337

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluzone High Dose Vaccine Then Fluzone High Dose Booster: Fluzone High dose vaccine administered at Day 0. Fluzone High dose vaccine administered as a booster after 30 days from the initial vaccine.
  Fluzone High Dose Vaccine
- Standard of Care: Fluzone High-Dose if age greater than or equal to 65 or Standard dose influenza vaccine if age less than 65 at day 0. Placebo administered 30 days after the initial vaccine.
  Standard of care/Placebo
Period: Overall Study
Arm/Group | Fluzone High Dose Vaccine Then Fluzone High Dose Booster | Standard of Care
Started (Initial Vaccine) | 81 | 41
Day 7 (+/- 2 Days) (Optional) (Research blood draw only) | 19 | 12
Day of Second Vaccine (30 Days After Initial Vaccine) | 74 | 41
30 Days Following 2nd Vaccine (30 Days After Second Vaccine) | 72 | 35
End of Study Visit (Optional) | 38 | 18
Completed (All Required Milestones) | 72 | 35
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone High Dose Vaccine Then Fluzone High Dose Booster | Standard of Care | Total
Number analyzed (Participants) | 81 | 41 | 122
Age, Continuous [Mean (Full Range); unit: years] | 67 [42 to 90] | 66 [37 to 89] | 67 [37 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 18 | 60
  Male | 39 | 23 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81 | 41 | 122
Detailed Diagnosis [Count of Participants; unit: Participants]
  Multiple Myeloma | 53 | 28 | 81
  WM | 6 | 4 | 10
  Other | 3 | 1 | 4
  Asymptomatic Myeloma | 8 | 1 | 9
  Asymptomatic WM | 0 | 3 | 3
  MGUS | 11 | 4 | 15
Disease Stage [Count of Participants; unit: Participants]
  Advanced | 64 | 32 | 96
  Early | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure by Primary Endpoint
Description: Any documented flu infection during the 2015-2016 flu season or evidence of disease progression.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone High Dose Vaccine Then Fluzone High Dose Booster | Standard of Care
Number analyzed (Participants) | 81 | 41
Participants | 26 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 12 months after initial vaccination
Description: The definition does not differ.
Arm/Group | Fluzone High Dose Vaccine Then Fluzone High Dose Booster | Standard of Care
All-Cause Mortality (participants affected / at risk) | 5/81 | 2/41
Serious Adverse Events (participants affected / at risk) | 8/81 | 1/41
Other Adverse Events (participants affected / at risk) | 0/81 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone High Dose Vaccine Then Fluzone High Dose Booster (N=81) | Standard of Care (N=41)
Intracranial hemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Immune system disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT02566265/Prot_SAP_000.pdf